CLINICAL TRIAL: NCT02801305
Title: Assessing and Comparing the Effect of Diltiazem Gel Versus Nitroglycerin Ointment in Healing Process of Scleroderma Digital Ulcers.
Brief Title: Diltiazem Gel Versus Nitroglycerin Ointment in Healing Process of Scleroderma Digital Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mohammad Ali Nazarinia (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Mohammad Ali Nazarinia, Associate Professor of Rheumatology, Shiraz University of Medical Sciences, Shiraz, Iran., Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 95010111653
Record Dates: First submitted 2016-06-09; First posted 2016-06-15 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Digital Ulcer of Scleroderma
Keywords: Scleroderma; Diltiazem; Nitroglycerin; Topical
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Nitroglycerin; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaseline (Placebo Comparator): About 60 patients will be considered to be in control group receiving vaseline ointment as the placebo applying 2 times daily on their ulcers for 8 weeks.
  Interventions: Drug: Vaseline
- Diltiazem Gel 2% (Experimental): About 30 patients will receive Diltiazem Gel 2% applying 2 times daily for 8 weeks on their digital ulcers.
  Interventions: Drug: Diltiazem Gel 2%
- Nitroglycerin Ointment 2% (Experimental): About 30 patients will receive nitroglycerin 2% applying 2 times daily for 8 weeks on their digital ulcers.
  Interventions: Drug: Nitroglycerin Ointment 2%

INTERVENTIONS:
Drug: Diltiazem Gel 2% — This a topical agent which will be applied on digital ulcers by scleroderma patients.
  Other Names: DILTIGEL
  Arms: Diltiazem Gel 2%
Drug: Nitroglycerin Ointment 2% — This a topical agent which will be applied on digital ulcers by scleroderma patients.
  Other Names: NITROCARD
  Arms: Nitroglycerin Ointment 2%
Drug: Vaseline — This is used as the topical placebo agent.
  Arms: Vaseline

SUMMARY:
Digital ulcers are one of the most prevalent complications of scleroderma (systemic sclerosis). There can be found few surveys on effect of topical agents on healing process of the ulcers. Thus, the aim of this study is to assess and compare the effects of topical diltiazem on SSc digital ulcers versus topical nitroglycerin.

DETAILED DESCRIPTION:
Introduction:

Systemic sclerosis, also named scleroderma (SSc), is an autoimmune connective tissue disease associated with small vessels vasculopathy and collagen deposition in skin and other internal organs [1, 2]. About 30-60 % of patients with limited and diffused type of scleroderma developed by digital ulcers (DUs) in course of their disease [3]. Depending on the sites of the ulcers, their pathophysiology is differed. The ones on distal parts of the digits are related to ischemic changes based on Raynaud phenomenon, intimal fibroproliferation, and thrombosis; while, the ones on bony prominences are mostly due to microtrauma and following poor vascularization for its healing [4].

These ulcers can affect the quality of life of the patients mostly due to the pain and difficulty in their healing [3]. Accordingly, several therapies have been introduced for improving its healing process. Among them, nitroglycerin ointment was assessed to be an effective topical agent on Raynaud phenomenon; however, there can be found only one study assessing its effect on SSc digital ulcer, which was shown to be non significant [5-7].

Calcium channel blockers (CCB) such as diltiazem are also being used for Raynaud phenomenon in scleroderma patients. Yet, some of their potential side effects such as peripheral edema, hypotension, and headache limit the up titration of these classes of drugs [8]. Moreover, their therapeutic effects on SSc digital ulcers are still being questionable. Only, one clinical trial assessed the effect of nifedipine on ulcer healing, which resulted in non-significant difference compared with placebo[7].

In addition to systemic form of CCBs, topical form of them such as diltiazem gel is also being available. Previous studies introduced this form of diltiazem as a vasodilator, mostly, for treatment of chronic anal fissure [9]. Comparing its effects with topical nitrate for chronic anal fissures showed some controversies. Some studies resulted in no significant difference between them; yet, the study by Ala et al, demonstrated that diltiazem gel has superiority to nitroglycerin ointment [10, 11]. Another survey, in spite of finding non- significant difference between these two agents in treatment of anal fissure, gave priority to diltiazem gel because of headache induced by nitroglycerin ointment [12].

As it can be inferred from previous studies, most of the medications used for scleroderma DU healing are drugs applied for Raynaud phenomenon. In spite of the determined therapeutic effects of such drugs on this phenomenon, their efficacy on healing of DUs is still being obscured. Furthermore, because of the complications of systemic therapies and limitation in their dose up titrating, topical agents are being preferred. However, there has not still found an effective topical therapy for DU of scleroderma patients.

The effect of topical diltiazem as a vasodilator agent in treatment of anal fissure brings to mind this idea that it may be also effective in healing of scleroderma DUs. In addition, comparing the effect of diltiazem gel and topical nitrate in anal fissures, generally, suggest the preference of the former. However, there can not be found any survey comparing the effects of these two topical vasodilators in treatment of DU. Thus, in this study, we aim to assess the effect of topical diltiazem on SSc digital ulcers and compare it by topical nitroglycerin.

Material and Method:

A single blind case control study will be done on 90 scleroderma patients registered in Tertiary Centers of rheumatology diseases of Shiraz University of Medical Sciences, Shiraz, Iran. (The sample size was estimated using the formula of n = (Zα/2+Zβ)2 * (p1(1-p1)+p2(1-p2)) / (p1-p2)2 [ Zα/2 is the critical value of the Normal distribution at α/2 (for a confidence level of 95%, α is 0.05 and the critical value is 1.96), Zβ is the critical value of the Normal distribution at β (for a power of 80%, β is 0.2 and the critical value is 0.84) and p1 and p2 are the expected sample proportions of the two groups]).

Inclusion Criteria:

The patients' scleroderma was diagnosed based on criteria of LeRoy[13]. The ones with ages between 20-70 years old will be entered into the study. They, all, should have at least one active digital ulcer.

Exclusion Criteria:

The cases with comorbid diseases such as diabetes, thyroid disease and cardiovascular diseases will be excluded from the survey. Moreover, the patients who are smoker, opium addict or alcohol abuser will also drop out of the study. In addition, the ones who received inhaled or oral prostanoid in last 3 months, phosphodiesterase inhibitors except for intermittent treatment of erectile dysfunction in last 1 month and the ones received antibiotics 2 weeks prior to the study will, also, be excluded. The baseline hepatic function test will be assessed and the cases with moderate to severe hepatic impairment or increase in aminotransferase levels more than 3 will also be excluded from the survey.

The study design:

The patients will be divided into 3 groups; one control group consisting of 30 cases, and two experimental groups with 30 patients in each of them. The control one (C) receiving Vaseline ointment as placebo, the experimental group 1 (E1) which will receive diltiazem gel (2%) applied on DUs two times daily and experimental group 2 (E2) treating by nitroglycerin ointment (2%) applied two times daily for 8 weeks.

The number of the DUs and the mean diameter of all DUs will be measured in 3 groups at the beginning and at the end of the study. Moreover, the site of the ulcers (fingertip, proximal interphalangeal joint (PIP), distal interphalangeal joint (DIP), metacarpophalangeal joint (MCP)) will be also taken into account and be submitted for each patient.

The number of new DUs developing during the study and the difference between mean diameters of them will be compared between 3 groups. In addition, the difference in mean of DUs in different sites will also be compared to see which site has more responsiveness to topical therapeutic agents used in this survey.

Ethical Issues:

Informed consent to the entire protocol as well as forms compatible with Helsinki Declaration was obtained from each patient. Ultimately, the ones who agreed to enroll will be recruited for the study.

Statistical Analysis:

Data will be entered into SPSS 19. For comparing the number and mean difference of digital ulcers' diameters between 3 groups and between different sites of the ulcer, one-way ANOVA will be applied. In addition, Bonferroni test as the post hoc of ANOVA will be applied for pairwise comparison of the groups. The significant p-value in all studies will be considered <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having the criteria of LeRoy.
* Having ages between 20-70 years old
* Having at least one active digital ulcer

Exclusion Criteria:

* Having co-morbid diseases such as diabetes, thyroid and cardiovascular diseases
* Being smoker, opium addict or alcohol abuser
* Ones received inhaled or oral prostanoid in last 3 months, phosphodiesterase inhibitors except for intermittent treatment of erectile dysfunction in last 1 month and the ones received antibiotics 2 weeks prior to the study
* The ones with moderate to severe hepatic impairment or increase in aminotransferase levels more than 3

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assessing the effect of topical diltiazem on scleroderma digital ulcers' healing process according to their site and comparing it with topical nitroglycerin | 10 months

SECONDARY OUTCOMES:
To see if there is any significant difference in mean diameters of scleroderma digital ulcers between patients receiving placebo and ones treated with diltiazem gel | 6 months
To see if the patients, receiving diltiazem gel, develop significantly less numbers of new ulcers during the study | 6 months
To see if there is any significant difference in mean diameters of scleroderma digital ulcers between patients receiving placebo and ones treated with nitroglycerin ointment | 6 months
To see if ones receiving nitroglycerin ointment develop significantly less numbers of new ulcers during the study | 6 months
To see if ones receiving diltiazem gel have difference in mean diameters of ulcers and numbers of new ones with group receiving nitroglycerin ointment | 6 months
To compare the difference in mean diameter of digital ulcers according to their site in each experimental group | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Nazarinia, M.D., Study Director — Shiraz Geriatric Research Center, Shiraz University of Medical Sciences, Shiraz, Iran
Locations (1):
- Rheumatology Reseach Center, Shiraz University of Medical Sciences, Shiraz, Iran., Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
The individual characteristic and information of the patients will be preserved by the researches and won't be released.

REFERENCES:
- [Background] Katsumoto TR, Whitfield ML, Connolly MK. The pathogenesis of systemic sclerosis. Annu Rev Pathol. 2011;6:509-37. doi: 10.1146/annurev-pathol-011110-130312. PMID 21090968
- [Background] Korn JH, Mayes M, Matucci Cerinic M, Rainisio M, Pope J, Hachulla E, Rich E, Carpentier P, Molitor J, Seibold JR, Hsu V, Guillevin L, Chatterjee S, Peter HH, Coppock J, Herrick A, Merkel PA, Simms R, Denton CP, Furst D, Nguyen N, Gaitonde M, Black C. Digital ulcers in systemic sclerosis: prevention by treatment with bosentan, an oral endothelin receptor antagonist. Arthritis Rheum. 2004 Dec;50(12):3985-93. doi: 10.1002/art.20676. PMID 15593188
- [Background] Ngcozana T, Ong V, Denton CP. Management of digital vasculopathy in systemic sclerosis: benefits of multiple courses of endothelin-1 receptor antagonists. BMJ Case Rep. 2014 Mar 28;2014:bcr2013203174. doi: 10.1136/bcr-2013-203174. PMID 24682137
- [Background] Herrick AL, Gush RJ, Tully M, Jayson MI. A controlled trial of the effect of topical glyceryl trinitrate on skin blood flow and skin elasticity in scleroderma. Ann Rheum Dis. 1994 Mar;53(3):212. doi: 10.1136/ard.53.3.212-a. No abstract available. PMID 8154944
- [Background] Abraham S, Steen V. Optimal management of digital ulcers in systemic sclerosis. Ther Clin Risk Manag. 2015 Jun 15;11:939-47. doi: 10.2147/TCRM.S82561. eCollection 2015. PMID 26109864
- [Background] LeRoy EC, Medsger TA Jr. Criteria for the classification of early systemic sclerosis. J Rheumatol. 2001 Jul;28(7):1573-6. PMID 11469464
- [Result] Anderson ME, Moore TL, Hollis S, Jayson MI, King TA, Herrick AL. Digital vascular response to topical glyceryl trinitrate, as measured by laser Doppler imaging, in primary Raynaud's phenomenon and systemic sclerosis. Rheumatology (Oxford). 2002 Mar;41(3):324-8. doi: 10.1093/rheumatology/41.3.324. PMID 11934971
- [Result] Tingey T, Shu J, Smuczek J, Pope J. Meta-analysis of healing and prevention of digital ulcers in systemic sclerosis. Arthritis Care Res (Hoboken). 2013 Sep;65(9):1460-71. doi: 10.1002/acr.22018. PMID 23554239
- [Result] Tsunoda A, Kashiwagura Y, Hirose K, Sasaki T, Kano N. Quality of life in patients with chronic anal fissure after topical treatment with diltiazem. World J Gastrointest Surg. 2012 Nov 27;4(11):251-5. doi: 10.4240/wjgs.v4.i11.251. PMID 23494072
- [Result] Bulus H, Varol N, Tas A, Coskun A. Comparison of topical isosorbide mononitrate, topical diltiazem, and their combination in the treatment of chronic anal fissure. Asian J Surg. 2013 Oct;36(4):165-9. doi: 10.1016/j.asjsur.2013.01.010. Epub 2013 Mar 6. PMID 24054756
- [Result] Ala S, Saeedi M, Hadianamrei R, Ghorbanian A. Topical diltiazem vs. topical glyceril trinitrate in the treatment of chronic anal fissure: a prospective, randomized, double-blind trial. Acta Gastroenterol Belg. 2012 Dec;75(4):438-42. PMID 23402088